CLINICAL TRIAL: NCT03986021
Title: Reproductive Axis Maturation in the Early Post-Menarchal Years: A Pilot Study
Brief Title: Reproductive Axis Maturation in the Early Post-Menarchal Years
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190110; 19-E-0110
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Reproductive Physiological Processes; Pediatrics; Adolescent Health; Adolescent Development
Keywords: Menarche; Adolescent; Physiology; Hormones; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- At-risk girls: Girls with first degree relative diagnosed with Polycystic Ovary Syndrome (PCOS) age 8-<15
- early post-menarche girls: Healthy, early post-menarchal girls age 8-<15
- Healthy control women: Women age >18-34 without PCOS at least 3-years post-menarchal with regular menstrual cycles every 21-35 days
- late post-menarche girls: Late post-menarchal girls age 11-<17.5 (gynecological age 2-5)
- Mothers of pediatric study participants: Mothers age 18-65 whose daughter has provided at least one vaginal swab sample for the First Period study.
- pre-menarche girls: Healthy, pre-menarchal girls age 8-<14.5
- Women with PCOS: Women diagnosed with PCOS >18-34 at least 3-years post-menarchal with irregular menstrual cycles

SUMMARY:
Background:

Most adult women with irregular periods of unknown cause report symptoms dating back to early adolescence. This study aims to learn how girls' periods change in the 2 years after their first period. We are also looking at girls who may have a condition called PCOS. This will help researchers learn what healthy puberty looks like and how they can spot signs of hormone problems early on.

Objective:

To learn how long it takes girls to develop regular menstrual cycles after their first period.

Eligibility:

Healthy girls ages 8-14 who either (1) haven't had their first period but show signs of puberty, such as breast development and hair in the genital area; or (2) had their first period in the past 6 months

Girls at risk for PCOS age 8-14 who have a mom or sister with PCOS

Girls with irregular menstrual cycles age 11-17.5

To compare with the girls, we are looking at women >=18-34 years old with PCOS,

Healthy women >= 18-34 years old without PCOS,

and Mothers of pediatric participants age 18-65

Design:

Both parents or guardians must allow their daughter to participate. They must attend all study visits with her.

Participants will first be screened by phone. Those who qualify will be screened in person. They will have a physical exam. They will give blood and urine samples. They will have an ultrasound of their abdomen. They will fill out questionnaires. They will sit in a BOD POD for 6 minutes: This is an egg- shaped machine that takes body measurements. They have the option to provide DNA samples.

Participants will have sets of visits at home or at the clinic about every 6 months. The number of visits in each set will depend on their menstrual cycle. Then they will have a final visit. Visits will include repeats of the screening tests. There are additional parts that participants may choose to be involved in depending on how involved they want to be.

At home, participants will collect their urine daily to measure hormones. They will keep a diary of their periods.

Adults: Women with known PCOS will complete the same Screening Visit as the girls and will collect dried urine specimens at home for 8 weeks;

The Healthy control women group will complete the same Screening Visit as the girls and collect dried urine specimens at home for 2 menstrual cycles;

The Mothers of pediatric participants group will complete a Screening Visit (informed consent, urine pregnancy test) and collect vaginal swab specimens at home for 2 menstrual cycles (approx. 8 weeks).

DETAILED DESCRIPTION:
The broad goal of these studies is to determine the physiologic and pathophysiologic underpinnings of irregular menstrual cycles among adolescents in general and those with increased genetic risk for polycystic ovarian syndrome (PCOS) in the early postmenarchal

period. Irregular menstruation affects > 2.5 million reproductive-age women in the US each year1. Most adult women with oligomenorrhea of unknown etiology reporting symptoms dating back to early adolescence. Importantly, irregular menstrual cycles during the teenage years may be a harbinger of future health risks extending beyond the reproductive system; among the nearly 80,000 female participants the Nurses' Health Study II, those with irregular and long cycles during adolescence and adulthood had a greater risk of premature mortality, particularly related to cardiovascular disease. While a period of cycle irregularity is well-described in the first few years after menarche, a lack of understanding of the basic mechanisms of normal reproductive axis development in the post-menarchal female has hampered our ability to distinguish abnormal from normal developmental trajectories. Moreover, the commonly held belief that menstrual irregularity among teenage girls is normal has also delayed detection of pathology in reproductive development, precluding institution of early preventative strategies to curtail future reproductive morbidity.

ELIGIBILITY:
* Part 1 - Pre-menarche monitoring ("holding pattern"):

Inclusion Criteria:

* Age 8-14.5 years old
* Healthy weight, defined as having a body weight >85% of expected (EBW) and a body mass index (BMI) <99th percentile
* Some breast development
* Pre-menarche

Exclusion Criteria:

* Taking or planning to take medications that affect reproductive hormones in the next 2 to 3 years (e.g. birth control pills, biotin supplements).
* Planning to move more than 60 miles from the CRU within the next 2 to 3 years
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* First-degree relative with polycystic ovarian syndrome, premature ovarian insufficiency, hypogonadotropic hypogonadism, or other pubertal development disorder
* Excessive exercise (defined as running >20 miles per week or its equivalent)
* Pregnancy

Part 2 - Post-menarche cycle tracking:

Inclusion Criteria:

* Age at menarche 10-14.5 years old
* Healthy weight, defined as having a body weight >85% of expected (EBW) and a body mass index (BMI) <99th percentile
* Approximately < 6 months post-menarchal (will typically have completed 4 or fewer menstrual cycles)
* Biochemical criteria: normal thyroid hormone, prolactin, and testosterone levels

Exclusion Criteria:

* Taking or planning to take medications that affect reproductive hormones in the next 2 to 3 years (e.g. birth control pills, biotin supplements).
* Planning to move more than 60 miles from the CRU within the next 2 to 3 years
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* First-degree relative with polycystic ovarian syndrome, premature ovarian insufficiency, hypogonadotropic hypogonadism, or other pubertal development disorder
* Excessive exercise (defined as running >20 miles per week or its equivalent)
* Anemia (defined as hemoglobin <12.0 g/dl)

  --Participants with hemoglobin between 11.5 g/dl and 12.0 g/dl may still participate by providing dried blood spots, or no more than 18 ml of blood during any given interval.
* Pregnancy

Part 3 - Intensive monitoring of ovarian follicle growth

Inclusion Criteria:

* Age at menarche 10-14.5 years old
* Healthy weight, defined as having a body weight >85% of expected (EBW) and a body mass index (BMI) <99th percentile
* Within 1 year of menarche
* Biochemical criteria: normal thyroid hormone, prolactin, and testosterone levels

Exclusion Criteria:

* Taking or planning to take medications that affect reproductive hormones in the next 1-2 years (e.g. birth control pills, biotin supplements).
* Planning to move more than 60 miles from the CRU within the next year
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* First-degree relative with polycystic ovarian syndrome, premature ovarian insufficiency, hypogonadotropic hypogonadism, or other pubertal development disorder
* Excessive exercise (defined as running >20 miles per week or its equivalent)
* Anemia (defined as hemoglobin <12.0 g/dl)

  --Participants with hemoglobin between 11.5 g/dl and 12.0 g/dl may still participate by providing dried blood spots, or no more than 18 ml of blood during any given interval.
* Pregnancy

Part 4 - Late Post-menarche cycle tracking:

Inclusion Criteria:

* Age 11-17.5 years old
* Approximately 2-5 years post-menarchal
* Biochemical criteria: normal thyroid hormone and prolactin

Exclusion Criteria:

* Taking or planning to take medications that affect reproductive hormones in the next 2 to 3 years (e.g. birth control pills, biotin supplements).
* Planning to move more than 60 miles from the CRU within the next 6 months
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* Anemia (defined as hemoglobin <12.0 g/dl)

  --Participants with hemoglobin between 11.5 g/dl and 12.0 g/dl may still participate by providing dried blood spots, or no more than 18 ml of blood during any given interval.
* Pregnancy

Adolescent girls, at-risk daughters, or sisters of women with PCOS

The girls with mothers or sisters with PCOS group will complete the Screening Visit and Parts 1-3. The same inclusion and exclusion criteria apply for Parts 1, 2, and 3 as stated above except that these individuals must have a first-degree relative with PCOS and they can have high androgen levels, excess body hair, and severe acne at screening.

Women with known PCOS (activities for 8 weeks only)

Inclusion Criteria:

* Age >=18-34 years old
* PCOS diagnosis
* at least 3-years post-menarchal with irregular menstrual cycles
* Biochemical (blood) or clinical signs of high androgen levels

Exclusion Criteria:

* Cannot be taking any medications that affect reproductive or metabolic hormones (e.g. birth control pill, biotin supplements, spironolactone, metformin).
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* Pregnancy

Healthy control women (Activities x 2 menstrual cycles)

Inclusion Criteria:

* Age >=18-34 years old
* at least 3-years post-menarchal with regular menstrual cycles every 21-35 days

Exclusion Criteria:

* Cannot be taking any medications that affect reproductive or metabolic hormones (e.g. birth control pill, biotin supplements, spironolactone, metformin).
* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* PCOS diagnosis or first-degree relative with disorder
* Pregnancy

Mothers of pediatric participants (Activities for 8 weeks / 2 menstrual cycles)

Inclusion Criteria:

* Age >=18-65 years old
* Biological mother of A Girl's First Period participant

Exclusion Criteria:

* Chronic medical condition, including but not limited to diabetes mellitus, congenital adrenal hyperplasia, cystic fibrosis, sickle cell disease, inflammatory bowel disease, juvenile rheumatoid arthritis, and lupus.
* Pregnancy

Ages: 8 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy early post-menarchal girls age 8-<15 years; PCOS women and girls with first degree relatives with PCOS; Healthy women 18-34 years; Late post-menarchal girls age 11-<17.5; healthy pre-menarchal girls age 8-<14.5; mothers of pediatric participants age 18-65
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
To determine the time from menarche to regular ovulatory cycles, defined as two consecutive ovulatory cycles in girls of variable genetic risk for PCOS | Defined as two consecutive ovulatory cycles with normal (10-14 day) luteal phase length during the first two post-menarchal years
  We hypothesize that the temporal sequence of reproductive maturation will consist of anovulatory cycles (representing a time of unopposed estrogen exposure), ovulatory cycles with a short luteal phase (estrogen with low progesterone exposure), and finally, ovulatory cycles with a normal luteal phase length (estrogen action fully counterbalanced by progesterone action)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie D Shaw, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-E-0110.html